CLINICAL TRIAL: NCT06164730
Title: Open-label, Phase 1b, Single Ascending Dose Study to Evaluate the Safety of VERVE-102 Administered to Patients With Heterozygous Familial Hypercholesterolemia or Premature Coronary Artery Disease Who Require Additional Lowering of Low-density Lipoprotein Cholesterol
Brief Title: A Study of VERVE-102 in Patients With Familial Hypercholesterolemia or Premature Coronary Artery Disease
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Verve Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VT-10201
Record Dates: First submitted 2023-12-01; First posted 2023-12-11 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Heterozygous Familial Hypercholesterolemia; Premature Coronary Heart Disease
Keywords: VERVE-102; Familial Hypercholesterolemia; Coronary Artery Disease; Dose Escalation; Gene Editing; Base Editing; heart-2
MeSH Terms: conditions — Hyperlipoproteinemia Type II; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Single ascending dose escalation/adaptive design.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (6):
- Cohort 1: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-102.
  Interventions: Drug: VERVE-102
- Cohort 2: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-102.
  Interventions: Drug: VERVE-102
- Cohort 3: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-102.
  Interventions: Drug: VERVE-102
- Cohort 4: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-102.
  Interventions: Drug: VERVE-102
- Cohort 5: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-102.
  Interventions: Drug: VERVE-102
- Cohort 6: Single Ascending Dose Escalation (Experimental): Participants will receive a single dose of VERVE-102.
  Interventions: Drug: VERVE-102

INTERVENTIONS:
Drug: VERVE-102 — Intravenous (IV) infusion

SUMMARY:
VT-10201 is an Open-label, Phase 1b, Single-ascending Dose Study That Will Evaluate the Safety of VERVE-102 Administered to Patients With Heterozygous Familial Hypercholesterolemia (HeFH) or Premature Coronary Artery Disease (CAD) Who Require Additional Lowering of LDL-C. VERVE-102 Uses Base-editing Technology Designed to Disrupt the Expression of the PCSK9 Gene in the Liver and Lower Circulating PCSK9 and LDL-C. This Study is Designed to Determine the Safety and Pharmacodynamic Profile of VERVE-102 in This Patient Population.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of HeFH or premature CAD

Exclusion Criteria:

* Homozygous familial hypercholesterolemia
* Active or history of chronic liver disease
* Current treatment with PCSK9 inhibitor or prior treatment within specified timeframe
* Clinically significant or abnormal laboratory values as defined by the protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Estimated)
Dates: Start 2024-04-30 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs) | up to Day 365

SECONDARY OUTCOMES:
Evaluation of maximum observed concentration (Cmax) | up to Day 365
Evaluation of time to maximum observed concentration (tmax) | up to Day 365
Evaluation of terminal elimination half-life (t1/2) | up to Day 365
Percent and absolute change from baseline in plasma PCSK9 concentration | up to Day 365
Percent and absolute change from baseline in LDL-C | up to Day 365

CONTACTS AND LOCATIONS:
Locations (18):
- United States (4):
  - Clinical Study Center, Dothan, Alabama
  - Clinical Study Center, High Point, North Carolina
  - Clinical Study Center, DeSoto, Texas
  - Clinical Study Center, Renton, Washington
- Australia (3):
  - Clinical Study Center, Adelaide
  - Clinical Study Center, Melbourne
  - Clinical Study Center, Sydney
- Canada (4):
  - Clinical Study Center, Chicoutimi
  - Clinical Study Center, Montreal
  - Clinical Study Center, Toronto
  - Clinical Study Center, Vancouver
- Clinical Study Center, Rehovot, Israel
- Clinical Study Center, Christchurch, New Zealand
- United Kingdom (5):
  - Clinical Study Center, Birmingham
  - Clinical Study Center, Edinburgh
  - Clinical Study Center, London
  - Clinical Study Center, Manchester
  - Clinical Study Center, Nottingham